CLINICAL TRIAL: NCT01650207
Title: Acupuncture for Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CCH-110410
Record Dates: First submitted 2012-07-12; First posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Shoulder Pain in Hemiplegic Side After Stroke
Keywords: electroacupuncture; TENS; shoulder disorder; hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Acupuncture Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- EA group (Experimental): To acupuncture the Juanyu (Li15) & Jugu (Li16) with sensation of de-qi, and then give 50 Hz electrical stimulation for 20 minutes.
  Interventions: Procedure: acupuncture
- TENS group (Experimental): The electrical patches were placed on the Juanyu (Li15) & Jugu (Li16) or Juanyu (Li15), Quchi (Li11), Shousanli (Li10) & Hegu (Li4), connected to a TENS apparatus and then give 50 Hz electrical stimulation for 20 minutes.
  Interventions: Procedure: TENS
- sham-acupuncutre (Sham Comparator): The Park's Sham Device were placed on the Juanyu (Li15) & Jugu (Li16).
  Interventions: Procedure: sham acupuncture

INTERVENTIONS:
Procedure: acupuncture — All participants were received regular rehabilitation program, and received different interventions.
  treatment frequency: 20 minutes per session, once daily, 5 times a week for 2 weeks
  Arms: EA group
Procedure: TENS
  Arms: TENS group
Procedure: sham acupuncture
  Arms: sham-acupuncutre

SUMMARY:
Shoulder pain has been reported to be one of the most common complications after stroke. Several factors have been related to shoulder pain after stroke such as paralysis, restricted range of motion in the shoulder, spasticity, sensory abnormalities, but the relationship between these factors and pain was not discussed.

The aim of this study is to identify the efficacy of electroacupuncture in reducing upper limbs spasticity and shoulder pain in stroke patients, and to evaluate the quality of life (QOL) for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Stroke within 6 months from onset
* Hemiplegia with shoulder pain (VAS > 2)

Exclusion Criteria:

* previous pathology of the shoulder or cardiac pacemaker, and cognition problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
shoulder pain degrees | 10 days after first intervention
  pain VAS in passive shoulder ROM

SECONDARY OUTCOMES:
shoulder ROM | 10 days after first intervention
  passive shoulder ROM (abduction, ER)

CONTACTS AND LOCATIONS:
Overall Officials: Tasen Wei, Principal Investigator — Physical Medical and Rehabilitation, Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Dawan, Changhua, Taiwan